CLINICAL TRIAL: NCT04990700
Title: Effect of Partial Rib Resection On the Control of Post-thoracotomy Pain: A Randomized Prospective Study
Brief Title: Effect of Partial Rib Resection On the Control of Post-thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, İsmail Dal, Principal Investigator, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: SiyamiErsek
Record Dates: First submitted 2021-07-16; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Pain, Postoperative; Iatrogenic Injury; Post-thoracotomy Pain Syndrome
Keywords: Post thoracotomy pain; Iatrogenic rib fracture; Thoracotomy; Partial rib resection
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Clinical data of intervention group and control groups will be compared
Who Masked: Participant
Masking Description: Patients do not know which study group they are in. The researchers know which group the patients are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Includes patients undergoing routine thoracotomy
- Intervention Group (Experimental): The group that will undergo 1 cm partial rib resection during thoracotomy.
  Interventions: Procedure: Partial rib resection

INTERVENTIONS:
Procedure: Partial rib resection — 1 cm partial rib resection during thoracotomy opening
  Arms: Intervention Group

SUMMARY:
The aim of this study is to evaluate the effect of partial rib resection in reducing acute post-thoracotomy pain

DETAILED DESCRIPTION:
It is known that severe post thoracotomy pain can be reduced by half with some strategies to prevent pain development. It was thought that partial rib resection would reduce intercostal tension and prevent an uncontrolled fracture. Thus, it is argued that post thoracotomy pain can be reduced. Partial rib resection is applied in clinical practice in selected patient groups. However, we could not find a clinical study on this subject in the English literature. The aim of this study is to determine whether partial rib resection has an effect on the control of thoracotomy pain.

Before the thoracotomy incision, simple randomization will be performed by flipping a coin.

Routine thoracotomy incision will be performed in the control group. In the intervention group, approximately 1 cm segment of the 6th rib will be excised with a rib scissors before the thorax retractor was placed.

Pericostal suture technique will be used in both groups at thoracotomy closure. Demographic information of the cases, preoperative respiratory function parameters, body mass index, Visual Analogue Scale scores, complications and analgesic doses will be recorded in the Case Report Form regularly.

ELIGIBILITY:
Inclusion Criteria:

* Participants who underwent thoracotomy in our clinic in 2019-2020
* Participants signing an informed consent form

Exclusion Criteria:

* Thoracic wall tumor
* Invasion of the thoracic wall by extrathoracic malignancy
* Pleural pathology
* History of previous rib fracture
* History of previous thoracotomy
* History of thoracic radiotherapy
* Emergency surgery
* Simultaneous incisions other than thoracotomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Postoperative visual analog scale scores | 7 days
  Min:1, Max:10 points, Higher scores mean worse outcome

SECONDARY OUTCOMES:
Iatrogenic rib fractures | During operation
  Yes or no
Administered analgesic doses | Up to 4 weeks
  Milligram
Duration of drainage | Up to 4 weeks
  Days
Length of hospital stay | Up to 4 weeks
  Days
Number of participants with postoperative bronchopulmonary complications | Up to 4 weeks
  Yes or no

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Dal, PhD, Principal Investigator — Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Locations (1):
- Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerner P. Postthoracotomy pain management problems. Anesthesiol Clin. 2008 Jun;26(2):355-67, vii. doi: 10.1016/j.anclin.2008.01.007. PMID 18456219
- [Background] Meyers JR, Lembeck L, O'Kane H, Baue AE. Changes in functional residual capacity of the lung after operation. Arch Surg. 1975 May;110(5):576-83. doi: 10.1001/archsurg.1975.01360110122020. PMID 1093513
- [Background] Katz J, Jackson M, Kavanagh BP, Sandler AN. Acute pain after thoracic surgery predicts long-term post-thoracotomy pain. Clin J Pain. 1996 Mar;12(1):50-5. doi: 10.1097/00002508-199603000-00009. PMID 8722735
- [Background] Soto RG, Fu ES. Acute pain management for patients undergoing thoracotomy. Ann Thorac Surg. 2003 Apr;75(4):1349-57. doi: 10.1016/s0003-4975(02)04647-7. PMID 12683601
- [Background] Wu N, Yan S, Wang X, Lv C, Wang J, Zheng Q, Feng Y, Yang Y. A prospective, single-blind randomised study on the effect of intercostal nerve protection on early post-thoracotomy pain relief. Eur J Cardiothorac Surg. 2010 Apr;37(4):840-5. doi: 10.1016/j.ejcts.2009.11.004. Epub 2009 Dec 1. PMID 19954996
- [Background] El-Hag-Aly MA, Hagag MG, Allam HK. If post-thoracotomy pain is the target, Integrated Thoracotomy is the choice. Gen Thorac Cardiovasc Surg. 2019 Nov;67(11):955-961. doi: 10.1007/s11748-019-01126-2. Epub 2019 Apr 16. PMID 30993532